CLINICAL TRIAL: NCT04902482
Title: Recovery of Function Through Cycling Therapy With Virtual Reality Biofeedback in Chronically Spinal Cord-injured People
Brief Title: iCycle II: Recovery of Function Through FES Cycling With VR Biofeedback in People With SCI.
Acronym: iCycle
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 140131
Record Dates: First submitted 2021-05-07; First posted 2021-05-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Spinal Cord Injuries
Keywords: Rehabilitation; FES cycling; Virtual Reality; Biofeedback; Motor Function
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iCycle training (Experimental): Participants will attend 3 training sessions per week at the RNOH. During these sessions, participants will tether their wheelchair (from under the seat) to the front of the iCycle, and their feet will be attached to the iCycle pedals. For training, participants will complete virtual reality cycle races displayed on a large screen in front of the iCycle: the more voluntary effort the participant contributes the greater the speed of the avatar. During cycling, a motor will control cycling speed, and muscle stimulation (FES) will be applied to the leg muscles (right and left gluteus, quadriceps and hamstrings) on alternative revolutions of the pedals. A dashboard screen will display controls for the stimulation, speed, brake, game switch and an emergency stop. Sessions will increase from 20 mins or the maximum achievable at the start (whichever is lower) up to at least 1 hour.
  Interventions: Device: iCycle Mark 3

INTERVENTIONS:
Device: iCycle Mark 3 — The iCycle Mark 3 is a cycle ergometer, designed to be used by people with SCI while they are seated in their own wheelchairs. The purpose of iCycle is to stimulate the leg muscles in the correct phase for cycling while motivating the person with a Virtual Reality cycling event, perhaps a race, to try to use their muscles.

SUMMARY:
The annual incidence of traumatic spinal cord injury (SCI) is estimated at 2,500 (35 per week) in the UK and, due to advances in research and clinical management, the majority now have incomplete injuries, with significant potential for neurological improvement. Discovering ways to provide intensive, but cost-effective SCI rehabilitation is therefore increasingly important.

The iCycle combines functional electrical stimulation (FES) cycling with VR cycle-racing feedback, where winning correlates with voluntary effort, to promote recovery. The aim is to improve walking in people with incomplete injuries, fundamental to independence and quality of life as well as long-term health. More intensive rehabilitative training is associated with better outcomes: the iCycle has the potential to increase intensity of exercise without additional demands on therapists' time and therefore cost.

Following the encouraging results in an initial study; it is now important to find out whether recovery will continue at a similar rate if iCycle training continues beyond 4 weeks. Six volunteers with SCI will be recruited to participate in this 20 week, single-site open feasibility trial. The trial consists of an intervention phase lasting up to 12 weeks (3 iCycle sessions per week), and an 8-week follow-up phase. Outcome measures (ISNC-SCI motor scoring, Trunk Impairment scale, Walking Index for Spinal Cord Injury, 6-minute walk test, Goal Attainment Scale and TMS) will be taken every 4 weeks. The 12-week intervention phase will be separated into three 4-week blocks; at the end of each block participants may decide whether or not they wish to continue training.

DETAILED DESCRIPTION:
Recruitment:

Participants will be recruited from London Spinal Cord injuries Centre (LSCIC) at the Royal National Orthopaedic Hospital (RNOH) where the training intervention will be carried out. The study will also be advertised via relevant newsletters, bulletin boards, websites and mailing lists.

For each recruited participant, the study will be conducted for up to 20 weeks in total*. This includes: an intervention phase lasting up to 12 weeks and an 8-week follow-up phase. Outcome measure (OM) assessments will be carried out every 4 weeks (OM1-6) to collect study variables. OM assessments will be conducted by either the researcher or physiotherapist. Each OM assessment session will be broken into two parts, each lasting 2 hours.

* At the end of each 4-week block in the intervention phase, participants will be given the option to continue training for the next 4-week block, or to stop training.

Intervention Phase:

Visit 1: During first outcome measure visit (OM1), participants will attend the Aspire Create labs at the RNOH in Stanmore, where they will be given the opportunity to ask questions about the study, informed consent to participate in the study will be taken and demographic information recorded in the Case Report Form (CRF).

Visits 2-38; 36 training sessions (3days/week) & 3 sessions Outcome measure assessments (OM 2-4) During the intervention phase, participants will attend 3 training sessions per week for up to 12 weeks (participants may opt to withdraw from training after 4 or 8 weeks and, if they choose to withdraw, will be advanced to the follow-up phase); each session will last from 20 mins-1 hour depending on the maximum achievable endurance (plus an additional <30 mins for set-up in iCycle). Stimulation parameters will be recorded for each participant before training starts and a training diary will be completed during each training session.

During each training session

1. Electrodes will be placed on the quadriceps, hamstring and gluteal muscles.
2. Participants will be able to tether their wheelchair (from under the seat) to the front of the iCycle for security and hold the handlebars provided on the dashboard while cycling for further stability. These can be adjusted for comfort.
3. Muscle stimulation (FES) will be applied to the leg muscles on alternative revolutions of the pedals during a virtual reality cycle race(s). The more voluntary effort the greater the speed of the avatar.
4. Training will increase from 20 mins or the maximum achievable at the start (whichever is lower) up to at least 1 hour.

Outcome measures (OM 2-4) will be performed every 4 weeks during the intervention phase (on a separate day to training sessions). The same outcome measures conducted in the baseline phase are repeated here with the addition of an audio recorded interview conducted in the OM4 appointment.

Follow-up Phase:

Visits 39-40 - 2 sessions Outcome measures (OM 5-6) Following termination of training, no further intervention will be given. Outcome measure assessments (OM 5-6) will be performed every 4 weeks during the 8-week follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* Incomplete SCI above T12
* >12 months post injury
* Respond to FES
* No deteriorating condition or other co-morbidity that would make participation impractical or unsafe.
* Marginal walker defined as able to rise from a chair, stand for 10 seconds and walk >10 steps without human help (but may use an aid including parallel bars).

Exclusion Criteria:

* Cardiac pacemaker
* Pressure sores/skin problems
* Unhealed lower limb fractures
* Pregnancy
* Active heterotrophic ossification - lower limbs
* Severe osteoporosis
* Complex regional pain syndrome
* Implanted metal work at electrode site (< 3/12)
* Lower Limb Malignancy
* T6 and below spinal malignancy
* Uncontrolled autonomic dysreflexia
* History of knee dislocation/subluxation
* Allergy to electrodes
* Cognitive difficulties - must be able to demonstrate an understanding of the iCycle and the virtual reality cycling game
* Severe spasticity - Ashworth scale 4 or 5 in any lower limb muscle groups
* Neurological degenerative diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2022-01-06 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in International Standards of Neurological Classification for SCI (ISNC-SCI) Motor score. | 15 minutes
  This is a is a clinician-administered scale used to classify the severity (completeness) of injury in individuals with SCI.

SECONDARY OUTCOMES:
Change in Trunk Impairment Scale (TIS) score | 15 minutes
  The TIS scores, on a range from 0 to 23, static and dynamic sitting balance as well as trunk co-ordination. It aims to score the quality of trunk movement and to be a guide for treatment.
Change in Walking Index for Spinal Cord Injury (WISCI II) score | 15 minutes
  Assessment index to assess ability of walking after SCI. This is quantified using rank ordering and dimension of impairment from most severe impairment (0) to least severe impairment (20) based on the use of devices, braces and physical assistance
change in 6-minute walk test (6MWT) distance | 15 minutes
  A submaximal exercise test that measures the distance walked over a span of 6 minutes
Threshold of evoked responses to Transcranial Magnetic Stimulation (TMS) | 60 minutes
  TMS is used to activate the motor cortex, and motor evoked potentials (MEPs) are measured in lower limb muscles using electromyography, Threshold to elicit MEPs is measured in each muscle.
Audio/transcribed feedback from participants from semi-structured interview | 30 minutes
  A semi-structured interview will be conducted to assess the participants experience in the trial, the training intervention and using the iCycle.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal National Orthopaedic Hospital, Stanmore, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: No
As the study is only 6 participants IPD will be provided in study publications.